CLINICAL TRIAL: NCT06150040
Title: A Phase I/II Study to Evaluate the Safety Clinical and Biological Activity of a Humanized Monoclonal Antibody Targeting Netrin-1 (NP137) in Combination With Standard AZACITIDINE+ VENETOCLAX in Patients With Refractory Acute Myeloid Leukemia
Brief Title: Acute Myeloid Leukemia Treated With With NETrin Abs in Combination With [AZACITIDINE + VENETOCLAX]
Acronym: AML-NET
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Centre Leon Berard (Other)
Collaborators: NETRIS Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET23-026; EU number (Other: 2023-503408-10-00)
Record Dates: First submitted 2023-11-10; First posted 2023-11-29 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia Refractory
Keywords: Acute Myeloid Leukemia; Unfit to intensive chemotherapy; NP137; Netrin-1; monoclonal antibody; Azacitidine and Venetoclax; Refractory to azacitidine and venetoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — netrin-1 inhibitor NP137; Azacitidine; venetoclax

STUDY DESIGN:
Intervention Model Description: The therapeutic combinations NP137 + [AZACITIDINE+VENETOCLAX] will be administered on the first 6 patients enrolled in the study at Dose Level (14 mg/kg). According to safety rules based on the dose limiting toxicities occurence, a dose reduction of NP137 at Dose Level -1 (9 mg/kg) will be assessed in 6 additional patients.
  After the safety run in part, study will be opened with 35 patients (including patients from the safety run in) at DL or DL-1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refractory Acute Myeloid Leukemia (Experimental): Patients who meet primary refractory disease definition according to ELN criteria after 2 cycles of standard [AZACITIDINE +VENETOCLAX] (i.e: patients who have failed to have a complete remission (with complete (CR) or incomplete hematologic recovery (CRi))
  Interventions: Drug: NP137; Drug: Azacitidine Injection; Drug: Venetoclax

INTERVENTIONS:
Drug: NP137 — IV infusion, 14mg/kg or 9mg/kg, every 2 weeks
Drug: Azacitidine Injection — Subcutaneous injection, 75 mg/m², on cycle Days 1-7 (28-days cycle)
Drug: Venetoclax — Orally, 70 mg, every day on Days 1-28

SUMMARY:
The aim of this study is to investigate the safety and the clinical activities of NP137 when combined with Azacitidine and Venetoclax in patients with refractory acute myeloid leukemia after 2 cycles of Azacitidine and Venetoclax.

DETAILED DESCRIPTION:
The dual treatment, VENETOCLAX and AZACITIDINE, is the standard of care for patients with newly diagnosed AML who are ineligible for intensive chemotherapy. However, upfront resistance as well as relapse following initial response demonstrate the need to improve this therapeutic strategy.

NP137 is a first-in-class humanized monoclonal antibody targeting specifically and selectively Netrin-1. Based on data collected from non clinical studies NP137 should act in synergy with VENETOCLAX and AZACITIDINE to reactivate and enhance the apoptotic pathway in AML cells.

The herein proposed study to assess the safety (Safety run in/ phase I part) and the preliminary efficacy signal (extension phase II part) of the NP137 when combined to AZACITIDINE AND VENETOCLAX in patients with refractory acute myeloid leukemia after 2 cycles of Azacitidine and Venetoclax.

This study will be an open-label, Phase I/II trial. the first part, consists to a safety run to assess the security and the tolerability of the drugs combination from the first 6 to 12 first patients enrolled into the study. All patients will receive a fixed dose of NP137 at the RP2D (Recommended Phase 2 Dose) determined from the First in human NP137 study(DL1) . A dose deescalation of NP137 is planned to DL-1 according to the Dose Limiting Toxicities observed during this period. The second part will be will be then conducted as a phase II using an adaptive Bayesian approach allowing to quickly stop treatment without evidence of efficacy. The clinical activity will be assessed based on ELN (European LeukemiaNet) criteria 2027 for the Acute Myeloid Leukemia.

ELIGIBILITY:
Inclusion Criteria:

I1. Adult is ≥ 65 years of age at the time of signing the ICF (Inform Consent Form)

I2. Histologically confirmed acute myeloid leukemia (AML) as defined by the 2022 World Health Organization (WHO) Classification.

I3. Patient previously untreated for AML (except with the first 2 cycles of his/her current A+V treatment) and who is considered as ineligible for induction regimen and intensive chemotherapy due to age and other comorbidity that the physician judges to be incompatible with such treatment:

OR Patient with expected poor prognosis under intensive /induction chemotherapy (e.g. with complex karyotype) OR "No-go" patients according ALFA decision tool ([e.i: patient with Adverse cytogenetics ≥1 of the following: mKRAS, mTP53)

Note : Patients with favourable-risk cytogenetics with intensive chemotherapy are not eligible, such as:

* t(8;21)(q22;q22.1); RUNX1-RUNX1T1
* inv(16)(p13.1q22) or t(16;16)(p13.1;q22); CBFB-MYH11
* Mutated NPM1 without FLT3-ITD or with FLT3-ITDlow†
* Biallelic mutated CEBPA

I4. Patients under treatment by A+V treatment as standard first line treatment for AML with no CR nor CRi after 2 cycles of AZACITIDINE +VENETOCLAX.

I5. Patient must be, in the judgment of the investigator, an appropriate candidate for an experimental therapy i.e. with no available other standard treatment or options except palliative care.

I6. Participant must have a life expectancy of at least 12 weeks.

I7. Participants has with Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 are eligible to the safety run-in part whatever their age. Then for the expansion part, patient with ECOG PS (Performance Status) of 0 to 2 for subject ≥ 75 years OR of 0 to 3 for subject ≥ 65 to 74 years of age are eligible.

I8. Demonstrate adequate cardiac function:

* QTc (corrected QT interval) ≤470ms
* Resting systolic BP <160mmHg
* Resting diastolic BP <100mmHg
* LVEF (left ventricular ejection fraction) ≥50% as determined by multiple-gated acquisition (MUGA) scan or transthoracic echocardiogram.

I9. Demonstrate adequate organ function as defined in table below, all screening laboratory tests should be performed within 7 days prior Cycle 1 day 1 :

* White Blood Cells Count < 25 × 109/L or lower; use of leukapheresis or hydroxyurea is permitted to achieve this concentration before Cycle 1 Day 1, at the discretion of the treating physician and according to institutional practice. (see exclusion criteria E6)
* Creatinine clearance Calculated creatinine clearance ≥30 mL/min determined by the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) formula OR via urine collection for 24-hour creatinine clearance or serum creatinine ≤ 2 upper limit of normal (ULN)
* Bilirubin Total bilirubin < 2 × the upper limit of normal (ULN) If total bilirubin ≥ 2 ULN, Direct Bilirubin must be < 2 x ULN unless considered due to leukemic organ involvement(< 5 ULN) and with the following Exception: Patients with known Gilbert disease who have serum bilirubin level ≤ 3 ULN may be enrolled.
* SGOT (serum glutamate oxaloacetate transaminase) (AST) and SGPT (serum glutamate pyruvate transaminase) (ALT) ≤ 3 x ULN unless considered due to leukemic organ involvement (< 5 ULN)

I10. Patient has no evidence of spontaneous tumor lysis syndrome (TLS) before NP137 introduction.

I11. Female subjects must be either:

* Postmenopausal; defined no menses for ≥ 12 months without an alternative medical cause; OR
* Permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)

I12. Non-sterile male subjects must use contraceptive methods with partner(s) prior to beginning study drug administration and continuing up to 3.5 months [106 days] after the last dose of NP137. Male subjects must agree to refrain from sperm donation from initial study drug administration during this same period.

I13. Patient must understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures.

I14. Patient must be able and willing to comply with study visits and procedures as per protocol.

I15. Patients must be covered by a medical insurance

Exclusion Criteria:

E1. Patient who is eligible for any curative therapy including but not limited to induction / intensive chemotherapies, CAR-T cell therapy and agrees to receive this therapy.

E2. Patient previously treated for AML with a hypomethylating agent and/or other chemotherapeutic agents either conventional or experimental for AML before NP137 introduction.

E3. Patient who has acute promyelocytic leukemia.

E4. Patient who experienced:

* Any persisting non hematological grade ≥ 3 AZACITIDINE AND VENETOCLAX related Adverse events before C1D1.
* Any vascular disorder grade ≥ 3 within 6 months prior C1D1.

E5. History of severe allergic anaphylactic reactions (≥ grade 3) to one of the components of the study drugs or to humanized antibodies or premedication and/or any of their excipients.

E6. Prior therapy or needs to be treated with a forbidden concomitant/concurrent therapies/procedures including:

* Any investigational agent or have used an investigational device.
* Major surgery within 4 weeks of start of study treatment. Participants must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment, C1D1.
* Anti-cancer treatment other than those specified in the protocol i.e. AZACITIDINE + VENETOCLAX.
* Live or live-attenuated vaccine within 30 days prior to the first dose of study treatments. Note: Inactivated vaccine are allowed.

Note:

* During the safety run in phase, Hydroxyurea is authorized prior C1D1 but a wash-out period of 2 days or 5*t1/2 before C1D1 whatever • shorter is required.
* During the expansion phase, the use of hydroxyurea for patients with rapidly proliferative disease is allowed during the course of cycle 1 at the discretion of the treating physician and according to institutional practice

E7. Active or untreated central nervous system involvement.

E8. Other invasive malignancy in the last 2 years except for those with a minimal risk of metastasis or death such as adequately managed in-situ carcinoma of the cervix, basal or squamous cell skin cancer, localized prostate cancer or ductal carcinoma in situ treated with curative intent, previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.

E9. Patients with any other known concurrent severe and/or uncontrolled medical condition including but not limited to diabetes, cardiovascular disease including hypertension, renal disease, or active uncontrolled infection, which could compromise participation in the study. For active infection requiring systemic therapy or fever likely secondary to infection within prior 48 hours: prophylactic antibiotics or prolonged course of IV antibiotics for controlled infection are allowed.

E10. Patients with uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure New York Heart Association (NYHA) class III/IV, clinically significant and uncontrolled arrhythmia as judged by the treating physician.

E11. Patient with evidence of uncontrolled active infection requiring systemic therapy (viral, bacterial or fungal).

E12. Patients known to be positive to HIV (testing will be performed a screening).

E13. Patients known to be positive for hepatitis B or C infection with the exception of those with an undetectable viral load within 3 months. Hepatitis B or C testing is not required and subjects with serologic evidence of prior vaccination to Hepatitis B virus (i.e., HBs Ag, anti-HBs+ and anti-HBc-) may participate.

Patients placed under a legal protection regimen: Judicial Safeguards, curatorship or guardianship.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Safety run in part : Incidence of Dose Limiting Toxicities (DLT) | 4 weeks
  To assess the safety of the proposed therapeutic combination [NP137 + AZACITIDINE VENETOCLAX] according to the incidence of Dose Limiting Toxicities (DLT) as defined per protocol.
Phase II part : Objective Response Rate (ORR) | 16 weeks
  To investigate the clinical activity of the proposed therapeutic combination [NP137 + AZACITIDINE + VENETOCLAX] through the Objective Response Rate (ORR) over the 4 cycles of AZACITIDNE +VENETOCLAX+ NP137 administration.
  ORR will be defined as the proportion of patients with a complete remission (CR) or complete remission with incomplete hematologic recovery (CRi), as best overall response over the 4 cycles of the study combination.

SECONDARY OUTCOMES:
Adverse events | from the date of first intake of study drug until to 90 days after study drug discontinuation, (at least up to 12 months for the last patient in)
  Incidence of any adverse events graded according to NCI-CTCAE V5.0
Duration of response | from the time of first documented response until the first progression or death, (at least up to 12 months for the last patient in)
  Measurement of the duration of response (CR/CRi)
Best overall response (BOR) | Every 28 days, up to 1 year
  Best overall response, is determined by the best response designation. For subjects without documented progression or subsequent anticancer therapy, all available response designations will contribute to the BOR determination :from the date of first intake of study drug until progression or at time of initiation of a new anti-cancer treatment
Objective Response Rate | 8 weeks
  Objective Response Rate after 2 cycles of study treatment defined as the proportion of participants who achieve: complete remission (CR) or complete remission with incomplete hematologic recovery (CRi) after 2 cycles of treatment (2 cycles of A+V including 4 injections of NP137)
Overall survival | Until up to 1 year follow-up of the last patient enrolled
  Overall survival measured from the date of treatment start to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Progression Free survival | Every 28 days, up to 1 year follow-up of the last patient enrolled
  Progression Free survival defined as the time from the initiation of the study treatment until first evidence of disease treatment failure : from the date of first intake of study drug until progression
Treatment Failure | Continuously, up to 1 year follow-up of the last patient enrolled
  Time to Treatment Failure Rate (TTF) defined as the time from the initiation of study treatment to its early discontinuation. Reasons for prematurely discontinuing treatment can include cancer progression but also adverse events, patient choice, or death.
Death in Medullary Aplasia | Every 28 days, up to 1 year follow-up of the last patient enrolled
  Death in Medullary Aplasia Rate based on cytological assessment: Deaths occurring ≥7 days following completion of initial treatment while cytopenic, with an aplastic or hypoplastic bone marrow obtained within 7 days of death, without evidence of persistent leukemia.
Neutrophil / platelet count recovery | Continuously, up to 1 year follow-up of the last patient enrolled
  Time to neutrophil / platelet count recovery (absolute neutrophil count (ANC) > 1 × 109/L (defined as neutrophil recovery) and platelet count > 100 × 109/L (defined as platelet recovery)).
Pharmacokinetic parameter: Cmax | Cycle 1 day 1, pre-dose; cycle 1 day 1, 3hours post-dose; cycle 1 day 2; cycle 1 day 7 or day 8; cycle 1 day 15, pre-dose; cycle 7 day 1, pre-dose; if Grade ≥3 infusion-related reaction and at the end of treatment visit (each cycle is 28 days)
  Plasma peak concentration
Pharmacokinetic parameter: tmax | Cycle 1 day 1, pre-dose; cycle 1 day 1, 3hours post-dose; cycle 1 day 2; cycle 1 day 7 or day 8; cycle 1 day 15, pre-dose; cycle 7 day 1, pre-dose; if Grade ≥3 infusion-related reaction and at the end of treatment visit (each cycle is 28 days)
  Time to reach the peak concentration
Pharmacokinetic parameter: AUCt (Area under the concentration-time) | Cycle 1 day 1, pre-dose; cycle 1 day 1, 3hours post-dose; cycle 1 day 2; cycle 1 day 7 or day 8; cycle 1 day 15, pre-dose; cycle 7 day 1, pre-dose; if Grade ≥3 infusion-related reaction and at the end of treatment visit (each cycle is 28 days)
  Area under the concentration-time curve from time zero to the last sample with the quantifiable concentration
Pharmacokinetic parameter: AUC∞ (Area under the concentration-time) | Cycle 1 day 1, pre-dose; cycle 1 day 1, 3hours post-dose; cycle 1 day 2; cycle 1 day 7 or day 8; cycle 1 day 15, pre-dose; cycle 7 day 1, pre-dose; if Grade ≥3 infusion-related reaction and at the end of treatment visit (each cycle is 28 days)
  Area under the concentration-time curve from time zero to infinity corresponding to the definite integral of a curve that describes the variation of a drug concentration in blood plasma as a function of time (drug exposure in plasma)
Pharmacokinetic parameter: CL (Clearance) | Cycle 1 day 1, pre-dose; cycle 1 day 1, 3hours post-dose; cycle 1 day 2; cycle 1 day 7 or day 8; cycle 1 day 15, pre-dose; cycle 7 day 1, pre-dose; if Grade ≥3 infusion-related reaction and at the end of treatment visit (each cycle is 28 days)
  Clearance: volume of plasma from which NP137 is completely removed per unit time.
Pharmacokinetic parameter: t1/2 | Cycle 1 day 1, pre-dose; cycle 1 day 1, 3hours post-dose; cycle 1 day 2; cycle 1 day 7 or day 8; cycle 1 day 15, pre-dose; cycle 7 day 1, pre-dose; if Grade ≥3 infusion-related reaction and at the end of treatment visit (each cycle is 28 days)
  Terminal elimination half-life: time required for the amount of NP137 in the body to decrease by half.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Léon Bérard, Lyon, France